CLINICAL TRIAL: NCT03191383
Title: An Observer-blind Study to Assess the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Investigational RSV Vaccine (GSK3003891A), in Healthy Pregnant Women and Infants Born to Vaccinated Mothers
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the GlaxoSmithKline (GSK) Biologicals' Respiratory Syncytial Virus (RSV) Investigational Vaccine (GSK3003891A) in Healthy Pregnant Women and Infants Born to Vaccinated Mothers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was canceled due to instability of the PreF antigen during manufacturing. No safety concern has been identified in past or ongoing studies.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 204810; 2016-002733-30 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Maternal immunization; Immunogenicity; Vaccines; Safety; Reactogenicity; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- GSK3003891A vaccine formulation 1 mother Group (Experimental): Subjects in this group will receive a single 30µg dose of the GSK3003891A investigational vaccine, by intramuscular injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: RSV vaccine (GSK3003891A) formulation 1
- GSK3003891A vaccine formulation 2 mother Group (Experimental): Subjects in this group will receive a single 60µg dose of the GSK3003891A investigational vaccine, by intramuscular injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: RSV vaccine (GSK3003891A) formulation 2
- GSK3003891A vaccine formulation 3 mother Group (Experimental): Subjects in this group will receive a single 120µg dose of the GSK3003891A investigational vaccine, by intramuscular injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: RSV vaccine (GSK3003891A) formulation 3
- Control group (Placebo Comparator): Subjects in this group will receive a single placebo injection, intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Drug: Placebo (Formulation buffer S9b)
- GSK3003891A vaccine formulation 1 infant Group (No Intervention): Infants born to mothers vaccinated with a single 30µg dose of the investigational GSK3003891A vaccine
- GSK3003891A vaccine formulation 2 infant Group (No Intervention): Infants born to mothers vaccinated with a single 60µg dose of the investigational GSK3003891A vaccine
- GSK3003891A vaccine formulation 3 infant Group (No Intervention): Infants born to mothers vaccinated with a single 120µg dose of the investigational GSK3003891A vaccine
- Control infant Group (No Intervention): Infants born to mothers who received a single placebo injection

INTERVENTIONS:
Biological: RSV vaccine (GSK3003891A) formulation 1 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: GSK3003891A vaccine formulation 1 mother Group
Biological: RSV vaccine (GSK3003891A) formulation 2 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: GSK3003891A vaccine formulation 2 mother Group
Biological: RSV vaccine (GSK3003891A) formulation 3 — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: GSK3003891A vaccine formulation 3 mother Group
Drug: Placebo (Formulation buffer S9b) — Single dose administered intramuscularly at Day 0 in the deltoid region of the non-dominant arm
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of the investigational GSK RSV vaccine in pregnant women aged 18 to 40 years and infants born to the vaccinated women

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent for study participation of the mother obtained from the mother or the mother and father, as applicable by local law, prior to performance of any study specific procedure.
* Written informed consent for study participation of the infant obtained from the infant's mother and/or father, as applicable by local law, or legally acceptable representative [LAR] prior to performance of any study specific procedure.
* Subjects between, and including, 18 and 40 years of age at the time of the first study visit.
* Pregnant females > 24 weeks of gestation at the time of screening and at 28 0/7 to 33 6/7 weeks of gestation at the time of vaccination, as established by ultrasound examination and last menstrual period date.
* Healthy pregnant females as established by medical history and clinical examination before entering into the study.
* Pregnant females not at high risk for complications, as determined by the obstetrical risk assessment form.
* No significant foetal findings observed during a second or third trimester ultrasound.
* Subjects who are willing to provide cord blood.
* Subjects who do not plan to give their child for adoption or place the child in care.

Inclusion Criteria infants:

• Re-signed written informed consent for study participation of the infant obtained from the infant's mother and/or father, as applicable by local law, or LAR.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before vaccination , or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before vaccination and ending at delivery with the exception of seasonal influenza vaccine and diphtheria, tetanus, pertussis/tetanus, diphtheria, pertussis [dTpa/Tdap] vaccine as part of standard of care which may be administered ≥ 15 days before or after study vaccination.
* Chronic administration of systemic immunosuppressants or other immune-modifying drugs, as well as administration of long-acting immune-modifying drugs during the period starting 6 months prior to study vaccination, or planned administration up to delivery. Topical steroids are allowed. Inhaled steroids are allowed up to the limit of ≤500 µg/day for beclomethasone or fluticasone, or ≤ 800 µg/day for budesonide.
* Administration of immunoglobulins (with the exception of prophylactic anti-Rh0D immune globulin) and/or any blood products during the period starting 3 months before study vaccination or planned administration during the study period.
* Previous experimental vaccination against RSV.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Low lying placenta during the current pregnancy, unless there is documented sonographic evidence that the placenta has moved up prior to enrolment.
* Any abnormal finding observed in nuchal translucency scan, serum testing and any other prenatal tests, if conducted.
* Incompetent cervix or cerclage during the current pregnancy.
* Having received medical treatment for suspected preterm delivery during the current pregnancy.
* Prior preterm delivery or having ongoing intervention in current pregnancy to prevent preterm delivery.
* Prior stillbirth or neonatal death, or ≥ 2 spontaneous abortions.
* Personal history of major congenital anomalies or early onset of eclampsia/pre-eclampsia in previous pregnancy.
* 1st degree relatives family history of major congenital anomalies and/ or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hemodynamically significant cardiac disorders.
* Gestational diabetes as determined by glucose challenge/tolerance test conducted after 20 weeks of gestation or as per local recommendations of the country, requiring intervention other than diet for control. In countries where glucose challenge/tolerance testing is not routinely performed in all pregnant women, should the screening urinalysis test show presence of glucose in urine, a glucose challenge/tolerance test should be performed and results should be available prior to enrolment, in order to exclude gestational diabetes prior to subject receiving the study vaccine.
* History of gestational diabetes in previous pregnancy(ies).
* Hypertension during the current pregnancy as defined below or if any antihypertensive medication is being provided, or history of hypertension requiring antihypertensive medication:

Hypertension during current pregnancy is defined as:

* a blood pressure systolic > 140 and/or diastolic 90 mmHg, documented in at least 2 separate measurements .

  * Current obstetric cholestasis or history of obstetric cholestasis.
  * Asthma and/or chronic obstructive pulmonary disease [COPD] if the subject is receiving treatment with chronic systemic glucocorticoids at any dose or inhaled glucocorticoids > 500 µg/day of beclomethasone or fluticasone, or > 800 µg/day of budesonide.
  * Significant neuro-psychiatric illness deemed likely to interfere with protocol compliance, safety reporting or receipt of pre-natal care, or requiring treatment with psychotropic drugs.
  * Diagnosed with Zika virus infection or suspected to have or have had Zika virus infection during the current pregnancy.
  * Known HIV infection, as assessed by local standard of care serologic tests conducted during the current pregnancy and prior to enrolment.
  * Known or suspected Hepatitis B virus [HBV] or Hepatitis C virus [HCV] infection.
  * Known infection during the current pregnancy with Toxoplasma, Parvovirus B19, Syphilis, Rubella, cytomegalovirus [CMV] or primary Herpes Simplex.
  * Known foetal anomalies in the current pregnancy.
  * Any clinically significant haematological and/or biochemical laboratory abnormality.
* Subjects with haematological/ biochemical values out of normal range which are expected to be temporary may be re-screened at a later date within the allowed time interval.

  • Acute disease and/or fever within 3 days prior to enrolment .
* Fever is defined as temperature ≥ 37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route.
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* For subjects with acute disease and/ or fever at the time of enrolment, Visit 1 may be scheduled at a later date within the allowed time interval and gestational age.

  * History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
  * Hypersensitivity to latex.
  * Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
  * History of drug or alcohol abuse within the past 2 years.
  * Any condition which, in the investigator's opinion, would increase the risks of study participation to the unborn infant.
  * Planned move to a location that will prohibit participating in the trial until study end.

Exclusion Criteria infants:

• Any condition which, in the investigator's opinion, would increase the risks of study participation to the infant.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited local adverse events (AEs) | During a 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days)
  Assessed solicited local symptoms are pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevents normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Number of subjects with solicited general AEs | During the 7-day follow-up period after vaccination (i.e. the day of vaccination and 6 subsequent days)
  Assessed solicited general symptoms are fatigue, fever [defined as oral/axillary/tympanic route temperature equal to or above 37.5 degrees Celsius (°C) or ≥ 38 °C for rectal route], gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain] and headache. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevents normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination
Number of subjects with unsolicited AEs | During a 30-day follow-up period after vaccination (i.e. the day of vaccination and 29 subsequent days)
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevents normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Number of subjects with haematological abnormalities | At Day 0
  Haematological laboratory abnormalities include haemoglobin level, white blood cell count [WBC], lymphocyte, neutrophil, eosinophil, platelet count, red blood cell count and mean corpuscular volume.
Number of subjects with haematological abnormalities | At Day 7
  Haematological laboratory abnormalities include haemoglobin level, white blood cell count [WBC], lymphocyte, neutrophil, eosinophil, platelet count, red blood cell count and mean corpuscular volume.
Number of subjects with biochemical abnormalities | At Day 0
  Biochemical laboratory abnormalities include alanine amino-transferase [ALT], aspartate amino-transferase [AST], creatinine and blood urea nitrogen.
Number of subjects with biochemical abnormalities | At Day 7
  Biochemical laboratory abnormalities include alanine amino-transferase [ALT], aspartate amino-transferase [AST], creatinine and blood urea nitrogen.
Number of subjects with any serious adverse events (SAEs) | From study start (Day 0) up to 6 months after delivery
  SAEs are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Number of infant subjects with any SAEs | From birth up to 6 months after birth
  SAEs are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Number of subjects with pregnancy outcomes | From study start (Day 0) up to delivery
  Pregnancy outcomes include live birth with no congenital anomalies, live birth with congenital anomalies, foetal death/still birth with no congenital anomalies, foetal death/still birth with congenital anomalies, elective/therapeutic termination with no congenital anomalies and elective/therapeutic termination with congenital anomalies.
Number of subjects with pregnancy-related AEs of specific interest | From study start (Day 0) up to delivery
  Pregnancy-related adverse events of specific interest include: gestational diabetes, gestational liver disease (including obstetric cholestasis and acute fatty liver of pregnancy), chorioamnionitis, labour protraction and arrest disorders, maternal sepsis, pregnancy-related hypertension, preterm premature rupture of membranes, premature labour, intrauterine growth restriction/poor foetal growth, pre-eclampsia and eclampsia, vaginal or intrauterine haemorrhage, medical conditions necessitating early delivery (induced labour or urgent C-section) (placenta abruption, uterine infection, oligohydramnios, etc), maternal death.
Number of infant subjects with AEs of specific interest | From birth up to 6 months after birth
  Infant-related AEs of specific interest include preterm birth, neonatal death, low birth weight and/or small for gestational age, neonatal sepsis, foetal/perinatal distress or asphyxia, failure to thrive/growth deficiency, congenital anomalies and neurodevelopmental delay.

SECONDARY OUTCOMES:
Number of infant subjects with SAEs | From birth and up to study end (Year 2)
  SAEs are defined as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Number of infant subjects with AEs potentially related to maternal vaccination | From birth up to study end (Year 2)
  Related infant AEs = AEs occurring in the infant assessed by the investigator as potentially related to the vaccination of the mother.
Number of infant subjects with neuro-developmental delays | At Year 1 and Year 2
  Infant subjects with Ages and Stages Questionnaires version 3 (ASQ-3) scores in the grey and black zones for any of the 5 developmental areas or domains (communication, gross motor skills, fine motor skills, problem solving and personal-social) :
  Grey zone (i.e. Monitoring zone) score means that the child's score falls ≥ 1 but <2 standard deviations below the mean score in any developmental area.
  Black zone (i.e. Referral zone) score means that the child's score falls below the cut-off (i.e. 2 standard deviations below the mean score) in any developmental area. Infant subjects scoring in the black zone in any of the 5 domains of the ASQ-3 will be referred for formal neurological evaluation
Number of infant subjects referred for formal neurological evaluation | At Year 1 and Year 2
  Neuro-developmental formal evaluation will be performed, for infants with ASQ3 black zone scores, using the Bayley Scale for Infant Development, Version III (BSID-III) or an equivalent.
Number of infant subjects with confirmed developmental delay | At Year 1 and Year 2
  Infants confirmed as having neuro-developmental delay following formal evaluation using the Bayley Scale for Infant Development, Version III (BSID-III) or an equivalent.
Neutralizing antibody titres against RSV-A, for all vaccinated mothers | At pre-vaccination (Day 0), Day 30 and Day 60 post vaccination and at delivery
  Titres will be expressed as geometric mean titres (GMTs)
Neutralizing antibody titres against RSV-B, for all vaccinated mothers | At pre-vaccination (Day 0), Day 30 and Day 60 post vaccination and at delivery
  Titres will be expressed as geometric mean titres (GMTs)
Palivizumab competing antibody (PCA) concentrations, for all vaccinated mothers. | At pre-vaccination (Day 0), Day 30 and Day 60 post-vaccination and at delivery
  Concentrations will be expressed as geometric mean concentrations (GMCs)
Neutralizing antibody titres against RSV-A, for all infants born to vaccinated mothers | At birth, at Month 3 and at Month 6
  Titres will be expressed as geometric mean titres (GMTs). Infants will be allocated to one of the 2 defined sub-cohorts (Month 3 or Month 6) and have the blood sample for immunogenicity obtained at the corresponding sub-cohort timepoint.
Neutralizing antibody titres against RSV-B, for all infants born to vaccinated mothers | At birth, at Month 3 and at Month 6
  Titres will be expressed as geometric mean titres (GMTs). Infants will be allocated to one of the 2 defined sub-cohorts (Month 3 or Month 6) and have the blood sample for immunogenicity obtained at the corresponding sub-cohort timepoint.
PCA concentrations, for all infants born to vaccinated mothers | At birth, at Month 3 and at Month 6
  Concentrations will be expressed as geometric mean concentrations (GMCs). Infants will be allocated to one of the 2 defined sub-cohorts (Month 3 or Month 6) and have the blood sample for immunogenicity obtained at the corresponding sub-cohort timepoint.
Number of infant subjects with lower respiratory tract infection (LRTI), severe LRTI and respiratory tract infection (RTI) with parental concern (according to the case definitions) associated with a respiratory syncytial virus (RSV) infection | From birth up to study end (Year 2)
  Occurrence of RSV-LRTI, severe RSV-LRTI, RSV-RTI with parental concern
Number of subjects (vaccinated mothers) with medically-attended (MA) RTI associated with an RSV infection | From Day 0 up to Month 6 post delivery
  Occurrence of RSV associated MA-RTI. A MA-RTI is defined as a visit of the mother to a health care professional for any respiratory symptom, including cough, sputum production and difficulty breathing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (3):
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Ellensburg, Washington
- Finland (2):
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
- Spain (7):
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through https://www.clinicalstudydatarequest.com/ following the timelines and process described on this site.